CLINICAL TRIAL: NCT02320084
Title: A Non-interventional Post Authorization Study (PASS) to Evaluate Long-term Safety of Orfadin Treatment in Hypertyrosinemia Type 1 (HT-1) Patients in Standard Care
Brief Title: Long Term Safety Study of Orfadin Treatment in HT-1 Patients in Standard Clinical Care
Acronym: OPAL
Status: Completed | Type: Observational
Sponsor: Swedish Orphan Biovitrum (Industry)
Responsible Party: Sponsor
Other Study IDs: Sobi.NTBC-005
Record Dates: First submitted 2014-10-23; First posted 2014-12-19 (Estimated); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Hereditary Tyrosinemia, Type I
Keywords: HT-1; Hereditary Tyrosinemia, Type I; hypertyrosinemia type 1; Orfadin; Long term safety; Hereditary Tyrosinemia Type 1
MeSH Terms: conditions — Tyrosinemias | interventions — nitisinone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- HT-1 patients on Orfadin treatment: HT-1 patients on Orfadin (nitisinone) treatment
  Interventions: Drug: Nitisinone

INTERVENTIONS:
Drug: Nitisinone — Nitisinone according to prescription
  Other Names: Orfadin

SUMMARY:
The purpose of this study is to look at the long term safety profile of Orfadin treatment in patients suffering from hereditary tyrosinemia type 1 (HT-1). Patients included in the study will use Orfadin according to normal clinical practice.

DETAILED DESCRIPTION:
The planned study is a non-interventional study that will look at the long-term safety of Orfadin treatment in patients suffering from hereditary tyrosinemia type 1. Orfadin will be used according to normal practice . There is an ongoing post-marketing surveillance (PMS) program to monitor hepatic, renal, hematological, neurological and ophthalmic status in all patients treated with Orfadin. The Committee for medicinal Products for Human Use (CHMP) has required this program and have looked at the data for approximately 400 patients and found the benefit-risk ratio to be positive. The present study (PASS) will replace the ongoing PMS. The transition of countries will be gradual; starting in 2013.The study will include HT-1 patients on Orfadin treatment in standard clinical care as well as newly diagnosed patients just starting with Orfadin treatment.

ELIGIBILITY:
Inclusion Criteria:

* All HT-1 patients receiving Orfadin treatment are eligible for entry.

Exclusion Criteria:

* No exclusion criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients receiving Orfadin is eligible for the study
Sampling Method: Non-Probability Sample
Enrollment: 315 (Actual)
Dates: Start 2013-09 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Occurrence of Adverse events related to hepatic function | from 2005
  Occurrence of Adverse events related to hepatic function
Occurrence of Adverse events related to renal function | from 2005
  Occurrence of Adverse events related to renal function
Occurrence of Adverse events related to Ophthalmological function | from 2005
  Occurrence of Adverse events related to Ophthalmological function
Occurrence of Adverse events related to hematological function | from 2005
  Occurrence of Adverse events related to hematological function
Occurrence of Adverse events related to cognitive developmental function | from 2005
  Occurrence of Adverse events related to cognitive developmental function

SECONDARY OUTCOMES:
Occurrence of death | from 2005
  Occurrence of death
Occurrence of liver transplantation | from 2005
  Occurrence of liver transplantation
Occurrence of other Adverse Events | from 2005
  Occurrence of Adverse Events other than those related to hepatic, renal, ophthalmic, hematological or cognitive functions
Occurrence of discontinuation of Orfadin treatment | from 2005
  Occurrence of discontinuation of Orfadin treatment

CONTACTS AND LOCATIONS:
Overall Officials: Study Physician, Study Director — Swedish Orphan Biovitrum
Locations (76):
- Austria (2):
  - Swedish Orphan Biovitrum Investigational Site, Innsbruck
  - Swedish Orphan Biovitrum Investigational Site, Vienna
- Belgium (5):
  - Swedish Orphan Biovitrum Investigational Site, Antwerp
  - Swedish Orphan Biovitrum Investigational Site, Brussels
  - Swedish Orphan Biovitrum Investigational Site, Leuven
  - Swedish Orphan Biovitrum Investigational Site, Montegnée
  - Swedish Orphan Biovitrum Investigational Site, Woluwe-Saint-Lambert
- Swedish Orphan Biovitrum Investigational Site, Prague, Czechia
- Swedish Orphan Biovitrum Investigational Site, Copenhagen, Denmark
- Finland (2):
  - Swedish Orphan Biovitrum Investigational Site, Tampere
  - Swedish Orphan Biovitrum Investigational Site, Turku
- France (7):
  - Swedish Orphan Biovitrum Investigational Site, Angers
  - Swedish Oprhan Biovitrum Investigational Site, Lille
  - Swedish Orphan Biovitrum Investigational Site, Lyon
  - Swedish Orphan Biovitrum Investigational Site, Nantes
  - Swedish Oprhan Biovitrum Investigational Site, Paris
  - Swedish Orphan Biovitrum Investigational Site, Paris
  - Swedish Orphan Biovitrum Investigational Site, Talence
- Germany (9):
  - Swedish Orphan Biovitrum Investigational Site, Düsseldorf
  - Swedish Orphan Biovitrum Investigational Site, Erlangen
  - Swedish Orphan Biovitrum Investigational Site, Freiburg im Breisgau
  - Swedish Orphan Biovitrum Investigational Site, Hanover
  - Swedish Orphan Biovitrum Investigational Site, Heidelberg
  - Swedish Orphan Biovitrum Investigational Site, Leipzig
  - Swedish Orphan Biovitrum Investigational Site, Magdeburg
  - Swedish Orphan Biovitrum Investigational Site, München
  - Swedish Orphan Biovitrum Investigational Site, Reutlingen
- Hungary (2):
  - Swedish Orphan Biovitrum Investigational Site, Budapest
  - Swedish Oprhan Biovitrum Investigational Site, Szeged
- Swedish Orphan Biovitrum Investigational Site, Dublin, Ireland
- Italy (10):
  - Swedish Orphan Biovitrum Investigational Site, Bari
  - Swedish Orphan Biovitrum Investigational Site, Catania
  - Swedish Orphan Biovitrum Investigational Site, Florence
  - Swedish Orphan Biovitrum Investigational Site, Milan
  - Swedish Orphan Biovitrum Investigational Site, Monza
  - Swedish Orphan Biovitrum Investigational Site, Napoli
  - Swedish Orphan Biovitrum Investigational Site, Padua
  - Swedish Orphan Biovitrum Investigational Site, Roma
  - Swedish Orphan Biovitrum Investigational Site, Saliceto
  - Swedish Orphan Biovitrum Investigational Site, Torino
- Netherlands (2):
  - Swedish Oprhan Biovitrum Investigational Site, Amsterdam
  - Swedish Orphan Biovitrum Investigational Site, Utrecht
- Norway (5):
  - Swedish Orphan Biovitrum Investigational Site, Fredrikstad
  - Swedish Orphan Biovitrum Investigational Site, Levanger
  - Swedish Oprhan Biovitrum Investigational Site, Oslo
  - Swedish Orphan Biovitrum Investigational Site, Oslo
  - Swedish Orphan Biovitrum Investigational Site, Tromsø
- Poland (2):
  - Swedish Oprhan Biovitrum Investigational Site, Warsaw
  - Swedish Orphan Biovitrum Investigational Site, Warsaw
- Swedish Orphan Biovitrum Investigational Site, Coimbra, Portugal
- Spain (15):
  - Swedish Orphan Biovitrum Investigational Site, Albacete
  - Swedish Orphan Biovitrum Investigational Site, Almería
  - Swedish Orphan Biovitrum Investigational Site, Badalona
  - Swedish Orphan Biovitrum Investigational Site, Barakaldo
  - Swedish Orphan Biovitrum Investigational Site, Barcelona
  - Swedish Orphan Biovitrum Investigational Site, Las Palmas de Gran Canaria
  - Swedish Oprhan Biovitrum Investigational Site, Madrid
  - Swedish Orphan Biovitrum Investigational Site, Madrid
  - Swedish Orphan Biovitrum Investigational Site, Málaga
  - Swedish Orphan Biovitrum Investigational Site, Mérida
  - Swedish Orphan Biovitrum Investigational Site, Murcia
  - Swedish Orphan Biovitrum Investigational Site, Pamplona
  - Swedish Orphan Biovitrum Investigational Site, Santiago
  - Swedish Orphan Biovitrum Investigational Site, Seville
  - Swedish Orphan Biovitrum Investigational Site, Valencia
- Sweden (4):
  - Swedish Orphan Biovitrum Investigational Site, Gothenburg
  - Swedish Orphan Biovitrum Investigational Site, Stockholm
  - Swedish Orphan Biovitrum Investigational Site, Umeå
  - Swedish Orphan Biovitrum Investigational Site, Uppsala
- United Kingdom (7):
  - Swedish Oprhan Biovitrum Investigational Site, Birmingham
  - Swedish Orphan Biovitrum Investigational Site, Bradford
  - Swedish Oprhan Biovitrum Investigational Site, London
  - Swedish Orphan Biovitrum Investigational Site, London
  - Swedish Oprhan Biovitrum Investigational Site, Manchester
  - Swedish Orphan Biovitrum Investigational Site, Manchester
  - Swedish Orphan Biovitrum Investigational Site, Sheffield

IPD SHARING:
Plan to Share IPD: Undecided
Discussions ongoing with regards to data sharing/registry.